CLINICAL TRIAL: NCT02607462
Title: Single Injection of Platelet-rich Plasma (PRP) to m. Gluteus Medius During Total Hip Arthroplasty Using Direct Lateral (Hardinge) Approach
Brief Title: PRP Therapy to m. Gluteus Medius During THA
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Satakunta Central Hospital (Other)
Responsible Party: Principal Investigator, Jussi Kosola, Resident, researcher, Satakunta Central Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PRP THA 092015
Record Dates: First submitted 2015-11-02; First posted 2015-11-18 (Estimated); Last update posted 2016-04-19 (Estimated); Status verified 2016-04

CONDITIONS: Hip Osteoarthritis
MeSH Terms: conditions — Osteoarthritis, Hip

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No

ARMS (2):
- PRP (Experimental): Platelet-rich plasma taken made from centrifuged venous blood.
  Interventions: Biological: PRP
- Saline (Placebo Comparator): Sodium chloride 0.9% used as placebo.
  Interventions: Other: Placebo

INTERVENTIONS:
Biological: PRP
  Arms: PRP
Other: Placebo
  Arms: Saline

SUMMARY:
Study purpose is to evaluate perioperative usefulness of Platelet-rich Plasma (PRP) in total hip arthroplasty (THA) surgery. The study is designed as a randomized double blinded study using saline as placebo. The measurement outcomes includes objective variables (MRI, dynamometer) as well as subjective measurements (Oxford Hip Score, Harris Hip Score).

Patients are assigned to two different groups, according to a randomization list. PRP (approximately 9ml from which 1ml is delivered to in-house laboratory for the measurement of platelet count) is obtained from venous blood and applied to m. gluteus medius during the closure of modified lateral approach (Hardinge).

Study participants are evaluated preoperatively by trained physiotherapist. After surgery, participants undergo clinical evaluation and imaged (MRI) at 3 and 12 months post-operative. In the same time points, strength, Harris Hip Score and Oxford Hip Score. At the end of the study, the nature of the injected substance is revealed to the patients.

ELIGIBILITY:
Inclusion Criteria:

* Clinically and radiology confirmed arthritis which treatment is total hip arthroplasty.

Exclusion Criteria:

* Revision surgery, insulin dependent diabetes and other endocrinology disease, smoking, use of per os cortisone, malignancy, rheumatoid arthritis, any autoimmune disease, alcoholist, previous fracture to hip, patients with diagnosed mental illness, absolute contraindications for MRI study

Ages: 60 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2015-11; Primary Completion 2017-10 (Estimated)

PRIMARY OUTCOMES:
The decrease of T2 weighted signaling between PRP and placebo group | Change from 3 months at 12 months
  Quantitative method of tissue healing

SECONDARY OUTCOMES:
Differences in Harris Hip Score points between PRP and placebo group | Change from 3 months at 12 months
  Quality method of post-operative healing
Comparison of hip abduction strengths between PRP and placebo group using dynamometer | Change from 3 months at 12 months
  Quantitive method of abduction strengths

CONTACTS AND LOCATIONS:
Locations (1):
- Satakunta Central Hospital, Pori, Finland

REFERENCES:
- [Derived] Aavikko A, Puhakka J, Haapala J, Kukkonen J, Makela K, Kosola J. Perioperative platelet rich plasma (PRP) in total hip arthroplasty through the Hardinge approach: protocol to study the effectiveness for gluteus medius healing. J Exp Orthop. 2018 Jun 19;5(1):23. doi: 10.1186/s40634-018-0127-7. PMID 29923073